CLINICAL TRIAL: NCT03637322
Title: Evaluation of Implementation of the Phoenix PrEP Access Project for Youth Aged 13-24
Brief Title: Evaluation of Implementation of the Phoenix PrEP (Pre-Exposure Prophylaxis) Access Project for Youth Aged 13-24
Status: Completed | Type: Observational
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 17-196
Record Dates: First submitted 2018-02-27; First posted 2018-08-20 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Unsafe Sex; IV Drug Usage
MeSH Terms: conditions — Unsafe Sex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate the implementation of a PrEP program for youth aged 13-24 in Phoenix, AZ. Numbers of youth who initiate PrEP, how long they continue with PrEP, and the barriers for youth who are trying to initiate and continue taking PrEP will be examined.

DETAILED DESCRIPTION:
This observational study will describe the barriers encountered and the benefits found as youth engage in a PrEP program, the Phoenix PrEP Access Project and as they participate in PrEP provided through standard medical care. This study does not investigate the safety, efficacy or other medical benefits of PrEP, but looks at the issues surrounding youth who are trying to access PrEP.

ELIGIBILITY:
Inclusion Criteria

* sexually active youth aged 13 through 24,
* at risk for contracting HIV,
* Negative for HIV as indicated by Negative Elisa and Western Blot (WB) or Negative 4th Generation test,
* weight greater than 35kg,
* offered PrEP to reduce the risk of contracting HIV.

Exclusion Criteria

* Unknown or Positive HIV status,
* Renal Impairment as indicated by elevated BUN or Creatinine, abnormal urinalysis,
* Active infection with Hepatitis B Virus,
* Taking other medications containing Emtricitabine, Tenofovir or tenofovir alafenamide(TAF) such as Atripla, Complera, Emtriva, Genvoya, Odefsey, Stribild, and Viread taking drugs containing lamivudine,
* taking Hepsera,
* clinical symptoms consistent with acute viral infection within the past month.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth aged 13 through 24 in the Phoenix area who are high risk for HIV infections because of unsafe sex practices and or IV drug use and have been offered PrEP as part of their standard medical care.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
PrEP Uptake | 3 years
  Uptake of PrEP offered to youth presenting for PrEP ages 13-24

CONTACTS AND LOCATIONS:
Overall Officials: Janice Piatt, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Bill Holt Clinic, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No